## **Cover Page for Statistical Analysis Plan**

Official Title: Culturally-targeted Communication to Promote SARS-CoV-2 Antibody Testing in

Saliva: Enabling Evaluation of Inflammatory Pathways in COVID-19 Racial

Disparities

NCT Number: NCT04957082

Date: May 28, 2024

## **Statistical Analysis Plan:**

The primary analysis for all study outcomes is based on assessing mean differences across the three study arms. Our arms include African Americans and Whites assigned to the general antibody testing video (groups 1 and 2) and African Americans assigned to the culturally-targeted video (group 3). A series of three-group one-way analysis of variance (ANOVAs) were conducted for all interval level/self-report outcomes, which included Theory of Planned Behavior and anticipatory racism measures. Planned comparisons were additionally conducted as LSD (non-alpha adjusted) two group comparisons. We also computed Cohen's d effect sizes to consider practical significance of pairwise differences.

For dichotomous (yes-no) outcomes related to accepting and completing the antibody test kit, we conducted chi square goodness of fit tests. We used planned two group comparisons to conduct follow-up analyses, which were also performed using chi square goodness of fit tests.

Please feel free to contact me at <a href="mailto:lucastod@msu.edu">lucastod@msu.edu</a> with any questions.

Thank you,

Todd Lucas, PhD
C.S. Mott Endowed Professor of Public Health
Charles Stewart Mott Department of Public Health
College of Human Medicine, Michigan State University